CLINICAL TRIAL: NCT03410472
Title: Assessing the Efficacy of Smart Phone Calorie Calculator Application on Body Composition With and Without Intervention
Brief Title: Assessing the Efficacy of Smartphone Calorie Calculator Application on Body Composition With and Without Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BHS-1309
Record Dates: First submitted 2017-11-16; First posted 2018-01-25 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: This is a randomized parallel design study
Who Masked: Outcomes Assessor
Masking Description: Only the individual performing the outcome measures will me masked to the assignment of the subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web based diet application (Experimental): This arm entails the subject to record their diet into an online web program to monitor calories. The calorie goal will be given to the subjects in this group prior to the study based on dual x-ray absorptiometry test that will test resting metabolic rate.
  Interventions: Behavioral: Web based diet application
- Control (No Intervention): This group will have body composition tested at week 1 and then repeat this test at 8 weeks having no intervention.

INTERVENTIONS:
Behavioral: Web based diet application — This group will be asked to record their diets for 8 weeks after being told an approximate calorie goal. This group will receive weekly emails with tips on how to eat healthy
  Arms: Web based diet application

SUMMARY:
Over nutrition has led to an increasing overweight and obese population. Maintaining a calorie deficit can be difficult causing many patients to be unsuccessful at weight loss attempts.

There are many smart phone applications that are labeled as weight loss aids, MyFitnessPal™ being one of these applications. MyFitnessPal ™ assists users to help record calorie intake to maintain a balanced caloric intake and to avoid over nutrition

Primary Hypothesis: This study is testing the hypothesis that subjects using a smart phone calorie calculator with intervention will have a greater body fat percentage loss in 8 weeks when compared to the control group.

Secondary Hypothesis: Subjects using a smart phone calorie calculator with intervention will report improved self-body image in 8 weeks.

DETAILED DESCRIPTION:
All subjects will read and sign an informed consent prior to participation in the study. The proposed study will be conducted at the Academic Health Care Center of the New York Institute of Technology, College of Osteopathic Medicine (Old Westbury, NY). Subjects will have 2 testing days where they will have to come into the Academic Health Care Center .

This study will consist of 30 participants and will last 8 weeks. Inclusion criteria will be male and female NYIT students between the ages of 18-35, a BMI ≥ 25.0, and own their own smart phone. All subjects will have their body composition measured, blood pressure, and pulse measured before and at the end of the study.

Participants will be randomly assigned by gender into two groups. Group one, the control group, will consist of 5 males, and 5 females. Group two, the intervention group, will consist of 10 males, and 10 females. At the start of the study both groups will have blood pressure, and pulse recorded, along with a duel x-ray absorptiometry body scan to measure resting metabolic rate (RMR) and body composition (lean body mass, body fat, BMI). At that time both groups will also receive the "NYC My Plate Planner", and the "USDA Dietary Guidelines for Americans 2015-2020".

Both Groups will be instructed to use the MyFitnessPal smart phone weight loss application to record calorie intake based on their resting metabolic rate determined by the body scan. Additionally both groups will initially receive a validated confidential survey on body image. The control group will not be contacted again until the end of the 8 weeks study. The intervention group will be contacted every week by email to discuss their weekly calorie intake, and compliance with the program. At week 4 each person in the intervention group will receive a phone call to discuss their calorie intake, and address any problems, or concerns. At the end of week 8 both groups will receive a follow up validated confidential survey on body image. At that time both groups will also return for a follow-up blood pressure recording, pulse recording, and body composition scan to measure resting metabolic rate and body composition (lean body mass, body fat, BMI).

ELIGIBILITY:
Inclusion Criteria:

* greater than 25 body mass index, must own a smart phone

Exclusion Criteria:

* currently using any other diet intervention

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2018-10-02 (Actual)

PRIMARY OUTCOMES:
Change in Body Fat Percentage | Week 1 and Week 8
  This will be tested using dual-x ray absorptiometry

SECONDARY OUTCOMES:
Change in Lean Body Mass | Week 1 and Week 8
  This will be tested using dual-x ray absorptiometry
Change in Body Mass Index | Week 1 and Week 8
  This will be tested using dual-x ray absorptiometry
Change in Systolic and Diastolic Blood Pressure | Week 1 and Week 8
  Blood pressure will be recorded using a manual sphygmometer
Change in BSQ-16 | Week 1 and Week 8
  This is a 16 question survey on body image

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Happel, DO, Principal Investigator — New York Institute of Technology College of Osteopathic Medicine
Locations (1):
- New York Institute of Technology, Old Westbury, New York, United States